CLINICAL TRIAL: NCT02232776
Title: A Prospective Study Evaluating the Efficacy and Safety of Losartan in Children With Immunoglobulin A Nephropathy
Brief Title: Efficacy and Safety of Losartan in Children With Ig A Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Losartan_IgA_2014
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2017-07

CONDITIONS: Glomerulonephritis, IGA
Keywords: Losartan; Ig A nephropathy; children; proteinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Losartan treatement (Experimental): All patients had received losartan treatment for 24 weeks.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — Dose of Losartan : 0.7mg/kg once daily.
  Other Names: Cozaar

SUMMARY:
The investigators hypothesize that using Losartan would help decrease proteinuria in controlling proteinuria in children with immunoglobulin A nephropathy.

DETAILED DESCRIPTION:
Twenty nine patient with IgA nephropathy with proteinuria (urine protein to creatinine ratio > 0.3 mg/mg) were included in the study. All patients had received losartan treatment for 24 weeks. Changes in blood pressure, proteinuria, renal function, and biochemical parameters were prospectively evaluated before and at 4 weeks and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2years or older and younger than 18 years
* Biopsy-proven Ig A Nephropathy
* Estimated GFR ≥ 90mL/min/m^2
* Mean urinary protein-creatinine ratio > 0.3 g/g from three first-morning spot urine collections

Exclusion Criteria:

* hypertension
* under dialysis or organ transplanted
* bilateral renal artery stenosis
* primary hyperaldosteronism
* pregnant

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
the change in urinary protein-creatinine ratio from baseline to the end of study | 24weeks
  Change in urinary protein excretion, determined as urinary protein-creatinine ratio compared to baseline, after 24 weeks of treatment.

SECONDARY OUTCOMES:
the change in urinary albumin-creatinine ratio from baseline to the end of study | 24 weeks
  Change in urinary albumin-creatinine ratio compared to baseline, after 24 weeks of treatment.
the proportion of patients wifh more than 50% decrease of urinary protein-creatinine ratio | 24 weeks
  Number of patients with wifh more than 50% decrease of urinary protein-creatinine ratio compared to baseline, after 24 weeks of treatment.
the proportion of patients wifh urinary protein-creatinine ratio < 0.2 at the end of study | 24 weeks
  Number of patients wifh urinary protein-creatinine ratio < 0.2 after 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Gyung Kang, Ph.D, Study Chair — Seoul National University Children's Hospital Departments of Pediatrics
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea